CLINICAL TRIAL: NCT01336764
Title: Enhancing Emotion Regulation During Driving in OEF/OIF Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Woodward, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WOS0016AGG
Record Dates: First submitted 2011-04-05; First posted 2011-04-18 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-04

CONDITIONS: Driving Distress Secondary to Trauma During Deployment
Keywords: driving distress; veterans; OEF/OIF

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Physical separation of Care Provider during self-administration of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): individual coping self-statements and stimulus guided paced breathing.
  Interventions: Behavioral: Cognitive reappraisal and breathing retraining
- Control (Sham Comparator): Coping self statements and breathing retraining will be replaced with undirected passive behaviors such as listening to music.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Cognitive reappraisal and breathing retraining — They will be induced to rapidly achieve reduced autonomic arousal through use of a graphics-rich biofeedback procedure and simultaneously engage in the generation and rehearsal of cognitive reappraisal scripts under the coaching of project therapist also in the vehicle.
  Arms: Active
Behavioral: Control — Unguided listening to radio/music.
  Arms: Control

SUMMARY:
Many U.S. military personnel are returning from Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) deployments with histories of trauma while driving in military vehicles. The proposed project aims to develop and test a rehabilitative technology aimed at enhancing emotion regulation and reducing operator-related risk during civilian driving.

DETAILED DESCRIPTION:
The driving exercises to be used are based upon standard Veterans Affairs-based driver assessments which have a well-established safety record and have been applied to a wide-range of medically-related and post-deployment driving issues.

Specifically, the driving exercises will embed a test-intervene-test session plan within a structured hierarchy of four progressively more challenging civilian driving tasks administered on successive weeks. Participants will drive local roads and highways familiar to Veterans Affairs - Palo Alto Health Care System Certified Driving Rehabilitation Specialists (CDRS). These courses have known characteristics as regards civilian driving challenges and OEF/OIF-relevant "trigger" stimuli. Graduation from one course to the next will take place only with permission from the CDRS who has accompanied the participant on the prior exercise. Based upon their self-reports of driving-related distress, we expect such distress to arise during the driving exercises. At such times, participants will be instructed to park in the next available safe parking location. They will be induced to rapidly achieve reduced autonomic arousal through use of a graphics-rich biofeedback procedure and simultaneously engage in the generation and rehearsal of cognitive reappraisal scripts under the coaching of project therapist also in the vehicle. These individualized procedures are expected to quickly lower emotional reactivity to subjectively adverse driving events and conditions. The participant will then drive the course a second time. Each session will finish with a graphical comparison of pre- and post-intervention vehicle and control surface movement parameters, visual attentional control, autonomic arousal and subjective driving distress.

ELIGIBILITY:
Inclusion Criteria:

1. Driving-related distress secondary to conditions of OEF/OIF deployment
2. Possesses valid driver's license
3. Owns vehicle registered in his/her name
4. Vehicle currently insured in his/her name
5. Drives regularly (e.g. to regularly scheduled activities such as work or school)
6. Drives to all driving rehabilitation appointments

Exclusion Criteria:

1. Any moving violations since discharge from the military
2. Any central nervous system injury or disease
3. Psychotic disorder and/or any psychotic signs or symptoms
4. Current alcohol or substance abuse/dependence (required answer: "yes" or "no", only)
5. Severe Post-traumatic Stress Disorder (as indicated by a PTSD Checklist (PCL) score greater than 60)
6. Severe Depression(as indicated by a Beck Depression Inventory-II score greater than 28)
7. Amputation or restricted mobility of any limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Woodward, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Control
Started | 12 | 10
Completed | 7 | 5
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Customized [Count of Participants; unit: Participants]
  age>/=18 years | 12 | 10 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Reduced Heart Rate During Driving (Aggregated Over Sessions)
Description: averaged over sessions
Time Frame: during 60-90 min driving intervention over the 3 intervention visits which were approximately one week apart
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Active | Control
Number analyzed (Participants) | 7 | 5
beats per minute | 3.21 (5) | 9.0 (5)

ADVERSE EVENTS:
Time Frame: Entire study
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 22/22
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No